CLINICAL TRIAL: NCT00115518
Title: Locoregional Radiotherapy in Combination With Cetuximab in Inoperable Non-Small Cell Lung Cancer Stage III
Brief Title: Radiation Plus Cetuximab in Locally Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Klaus Herfarth, MD, UJniversity of Heidelberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEAR L-284/2004
Record Dates: First submitted 2005-06-22; First posted 2005-06-23 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2011-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cetuximab — After Cetuximab loading dose. weekly cetuximab during RT. 13 weeks cetuximab weekly maintenance

SUMMARY:
The purpose of this trial is to study combined locoregional radiotherapy with cetuximab in non-operable NSCLC Stage III (Phase II trial).

Endpoints:

safety and feasibility (primary) response, survival, time to progression (secondary)

DETAILED DESCRIPTION:
Study entry examinations:

* blood cell count
* liver enzymes
* ventilatory function test
* pregnancy test (premenopausal women)
* CT of the thorax
* CT of the brain
* Ultrasound of the liver
* Bone scan
* FDG PET scan (after inclusion)

Follow-up examinations (2 months, than every 3 months):

* patients history and examination
* CT scan of the thorax
* ventilatory functions test
* FDG PET scan (at least at 6 months)
* bone scan (yearly)
* ultrasound of the liver (every 6 months)

Cetuximab administration:

* 450 mg / m^2 body surface on week 1
* 250 mg /m^2 body surface weekly, week 2 -21

Radiation therapy:

* intensity modulated radiation therapy of primary tumor and mediastinum (2 Gy single dose, total dose 50 Gy; 5 fractions per week) with boost to the PET positive sites (2 Gy single doses up to 66 Gy). Radiation therapy during weeks 2-8.

Amendment 1/07: 3D conformal RT possible, but not if FeV1 < 1.5L of < 50%

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified NSCLC
* Not eligible for Radiochemotherapy or patient refuses chemotherapy
* FeV1 >1.5 L or min. 50%
* KPI >= 70%
* Life expectancy > 6 months
* Weight loss less than 10% of body weight in 12 months
* Compliance
* Adequate blood counts (LC > 3000 x 10^3/ml, Tc >100000 x 10^3/ml, Hb > 10 g/dl)
* Effective contraception

Amendment 1/07: FeV1 >1.2 L or min 40%

Exclusion Criteria:

* Active infection
* Reduced liver function
* Vena cava superior syndrome
* Malignant pleural effusion
* Pregnancy or breast feeding
* Additional serious systemic disease
* Secondary malignancy (except carcinoma in situ of the cervix, basalioma of the skin, secondary cancer in remission for > 5 years)
* Known allergies against proteins
* History of former antibody therapy
* Allergy against i.v. contrast agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2009-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
safety: rate of side effects (skin reactions, allergic reactions, decrease of pulmonary function) | 3 yrs

SECONDARY OUTCOMES:
response (RECIST criteria of primary tumor and enlarged lymphnodes) | 3 yrs
survival (at 3 years) | 3 yrs
time to progression (locally and systemically) | 3 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Klaus K Herfarth, MD, Principal Investigator — Heidelberg University
Locations (1):
- University of Heidelberg, Heidelberg, Germany

REFERENCES:
- [Result] Jensen AD, Munter MW, Bischoff HG, Haselmann R, Haberkorn U, Huber PE, Thomas M, Debus J, Herfarth KK. Combined treatment of nonsmall cell lung cancer NSCLC stage III with intensity-modulated RT radiotherapy and cetuximab: the NEAR trial. Cancer. 2011 Jul 1;117(13):2986-94. doi: 10.1002/cncr.25888. Epub 2011 Jan 24. PMID 21264838
- [Derived] Jensen AD, Munter MW, Bischoff H, Haselmann R, Timke C, Krempien R, Sterzing F, Nill S, Heeger S, Hoess A, Haberkorn U, Huber PE, Steins M, Thomas M, Debus J, Herfarth KK. Treatment of non-small cell lung cancer with intensity-modulated radiation therapy in combination with cetuximab: the NEAR protocol (NCT00115518). BMC Cancer. 2006 May 8;6:122. doi: 10.1186/1471-2407-6-122. PMID 16681848